CLINICAL TRIAL: NCT01539213
Title: An Exploratory Study to Investigate the Distribution of Secukinumab (AIN457) Into Dermal Interstitial Fluid Using Open Flow Microperfusion After a Single Subcutaneous Administration of 300 mg in Healthy Subjects and Psoriatic Patients
Brief Title: Distribution of Secukinumab (AIN457) Into Dermal Interstitial Fluid After a Single Subcutaneous Administration of 300 mg
Acronym: OFM ISF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAIN457A2225; 2011-002929-21 (EudraCT Number)
Record Dates: First submitted 2011-12-23; First posted 2012-02-27 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2015-02

CONDITIONS: Healthy; Psoriasis
Keywords: Psoriasis; interstitial fluid; open flow microperfusion; IL-17; inflammatory skin disease; scaly patches; Healthy volunteers and psoriasis patients
MeSH Terms: conditions — Psoriasis; Dermatitis | interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AIN457 (Experimental): secukinumab (AIN457)
  Interventions: Drug: secukinumab (AIN457)

INTERVENTIONS:
Drug: secukinumab (AIN457) — anti-IL-17 antibody

SUMMARY:
The proposed exploratory study aims to understand the in vivo skin distribution properties of subcutaneously (s.c.) administered AIN457 in psoriatic and healthy skin using open flow microperfusion (OFM). The data of this study will help to understand the mode of action of AIN457 in its target tissue.

It aims to establish a technique assessing in vivo distribution of AIN457 and its metabolites in human dermal interstitial fluid (ISF) and exploring a potential pharmacodynamic effect in situ. In addition, the study will further evaluate safety and local tolerability of subcutaneously administered AIN457 and explore dermal interstitial fluid skin levels of potential disease relevant biomarkers.

The study is divided into two parts - Part I with 8 healthy volunteers (HV) to validate the method is completed and Part II with 8 psoriasis patients will start based on the outcome of Part I.

ELIGIBILITY:
For Part I : Healthy male and female subjects 18 to 65 years of age inclusive; For Part II: Chronic plaque-type psoriasis (with or without arthritis) diagnosed for at least 6 months before enrollment including at least one plaque accessible for OFM with at least moderate severity ; Key exclusion criteria for Part I and Part II: Women of child-bearing potential unwilling to use effective contraception; History of an ongoing, chronic or recurrent infectious disease, or evidence of tuberculosis infection as defined by a positive TB-test at screening; For Part I: Use of any prescription drugs, herbal supplements, within 4 weeks prior to initial dosing For Part II: Ongoing use of concomitant psoriasis treatments. Washout periods have to be adhered to.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Amount (ng/ml) of AIN457 in dermal interstitial fluid. | Day 8
  Distribution of AIN457 into dermal interstitial fluid after single subcutaneous administration of AIN457 in healthy subjects and in psoriatic patients
Amount (ng/ml) of AIN457 in dermal interstitial fluid. | Day 15
  Distribution of AIN457 into dermal interstitial fluid after single subcutaneous administration of AIN457 in healthy subjects and in psoriatic patients

SECONDARY OUTCOMES:
Number of adverse events to measure Safety of subcutaneously administered AIN457 in healthy volunteers and psoriatic patients | 3 weeks
  Safety of AIN457 s.c. injection will be documented as numbers of adverse event.
Part I only: concentration of sinistrin in serum vs. dermal interstitial fluid to confirm the ability of sinistrin to serve as reference to quantify AIN457 in dermal interstitial fluid. | Day 8
  Concentration of sinistrin in serum compared to dermal interstitial fluid.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Graz, Austria

REFERENCES:
- [Result] Abstracts of the 2013 International Investigative Dermatology Meeting. May 8-11, 2013. Edinburgh, Scotland, United Kingdom. J Invest Dermatol. 2013 May;133 Suppl 1:S1-311. No abstract available. PMID 23607128
- See also: Results for CAIN457A2225 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10883